CLINICAL TRIAL: NCT07154186
Title: Impact of Triglycerides Glucose Index on Angiographic Profiling of Non-Diabetic Premature Coronary Artery Disease Patients
Brief Title: Triglycerides Glucose Index on Angiographic Profiling of Non-Diabetic Premature Coronary Artery Disease Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Remon Saleh Adly, Lecturer of Cardiovascular, Faculty of Medicine, Sohag University, Sohag, Egypt., Sohag University
Other Study IDs: Soh-Med-25-5-5PD
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Triglycerides Glucose Index; Angiographic Profiling; Non-Diabetic; Premature; Coronary Artery Disease
MeSH Terms: conditions — Premature Birth; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group L: Patients with a low triglyceride-glucose (TyG) index tertile.
  Interventions: Other: Coronary Angiographic Assessment
- Group H: Patients with a high triglyceride-glucose (TyG) index tertile.
  Interventions: Other: Coronary Angiographic Assessment

INTERVENTIONS:
Other: Coronary Angiographic Assessment — Coronary angiographic assessment will be performed for all patients.

SUMMARY:
This study aims to evaluate the impact of the triglyceride-glucose (TyG) index on the angiographic profiling of non-diabetic patients with premature coronary artery disease (CAD).

DETAILED DESCRIPTION:
Premature coronary artery disease (CAD), defined as CAD occurring before the age of 55 in men and 65 in women, has emerged as a growing health concern worldwide.

Insulin resistance and associated metabolic alterations are strongly implicated in premature atherosclerosis. Even in non-diabetic individuals, subclinical insulin resistance promotes endothelial dysfunction, oxidative stress, and low-grade inflammation, leading to early vascular damage.

The triglyceride-glucose (TyG) index, calculated using fasting glucose and triglyceride levels, has emerged as a cost-effective surrogate marker for insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Non-diabetic patients [no history of diabetes, hemoglobin A1C (HbA1C) < 6.5%, fasting glucose < 126 mg/dL].
* Confirmed diagnosis of coronary artery disease (CAD) by coronary angiography.

Exclusion Criteria:

* Known diabetes mellitus (type 1 or type 2).
* Previous history of coronary revascularization.
* Severe hepatic or renal dysfunction [alanine transaminase (ALT)/aspartate aminotransferase (AST) ≥ 5× upper limit of normal (ULN), estimated glomerular filtration rate (eGFR)< 30 mL/min/1.73 m²].
* Malignant disease, autoimmune disease, or systemic inflammatory disorders.
* Current use of triglyceride-lowering medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study will be conducted at Sohag University Hospitals, following approval from the institutional ethics committee.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ischemia- driven revascularization | 6 months post-procedure
  Incidence of ischemia- driven revascularization will be recorded.

SECONDARY OUTCOMES:
Association between triglyceride-glucose index and single-vessel disease | 6 months post-procedure
  The association between the triglyceride-glucose (TyG) index and single-vessel disease (SVD) will be recorded.
Association between triglyceride-glucose index and two-vessel disease | 6 months post-procedure
  The association between the triglyceride-glucose index (TyG) and two-vessel disease (2VD) will be recorded.
Association between triglyceride-glucose index and three-vessel disease | 6 months post-procedure
  The association between the triglyceride-glucose index (TyG) and three-vessel disease (3VD) will be recorded.
Correlation of the triglyceride-glucose index with traditional cardiovascular risk factor | 6 months post-procedure
  Correlation of the triglyceride-glucose index with traditional cardiovascular risk factor will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.